CLINICAL TRIAL: NCT00346645
Title: A Phase II Study of Velcade® (Bortezomib) in Patients Stage IIIB OR IV Non-Small Cell Lung Cancer (NSCLC) Who Have Not Received Prior Chemotherapy
Brief Title: A Phase II Study of Velcade® in Patients Stage IIIB OR IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stopped after planned interim analysis for lack of efficacy
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VELCADE; CSET 1192
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2012-01

CONDITIONS: STAGE IIIB OR IV NON-SMALL CELL LUNG CANCER
Keywords: NON-SMALL CELL LUNG CANCER METASTATIC
MeSH Terms: interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomid (VELCADE®)

SUMMARY:
The purpose of this study is to determine whether Bortezomib is effective in the treatment of patients with non-small-cell lung cancer who have not received any prior chemotherapy regimen for advanced disease.

DETAILED DESCRIPTION:
Chemotherapy for non-small-cell lung cancer (NSCLC), mainly Cisplatin-based combinations, provides a measurable but modest survival benefit for selected patients with advanced disease. Advanced NSCLC remains largely fatal, with the positive impact of chemotherapy limited by intrinsic and acquired resistance, manifested clinically by early progression and transient responses. Current chemotherapy regimens have limited efficacy with a magnitude of survival benefit that is still modest, and lead to significant toxicity, with many patients unable to receive this kind of treatment, even in first line setting. There is, therefore, a great need to provide patients with less toxic agents such as the novel targeted therapies, with the potential to improve the efficacy and maintain a good quality of life. Bortezomib, a proteasome inhibitor, has shown benefit as single agent in pretreated patients with similar or lesser toxicity compared to chemotherapy. The current project is a phase II trial that will include 46 patients with advanced NSCLC and without prior chemotherapy. An early tumor assessment (after 6 weeks of therapy) will be performed, combined with regular clinical and symptom assessment to allow for rapid and appropriate management of non-responding patients, with cross over to another therapy as per the investigator and patient choice. The primary objective is efficacy of bortezomib as determined by the rate of no progression at 6 weeks. Secondary objectives are efficacy of bortezomib as determined by objective response rate (incidence of CR and PR), disease control rate (CR, PR and stabilization), duration of disease control, duration of objective response, progression-free survival,overall survival, safety of bortezomib, rate of doublet therapy in second line.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, inoperable, unresectable, incurable, locally advanced, recurrent or metastatic (Stage IIIB or Stage IV) non-small cell lung cancer. (Note: Histology is the preferred method of diagnosis. However, in case only cytology is available, specimens from brushing, washing or needle aspiration etc. are acceptable for diagnosis. Sputum cytology alone is not acceptable)
* No prior chemotherapy or therapy with systemic anti-tumour therapy (e.g., monoclonal antibody therapy). Prior surgery and/or localized irradiation (palliative RT or curative RT) is permitted. Pre operative or post operative anti neo-plastic therapy is allowed if ended more than 2 years ago
* No prior exposure to agents directed at the HER axis (e.g. EGFR TK Inhibitors, Herceptin)
* Measurable disease as defined by RECIST criteria (attachment 1)
* Age 18 or greater
* ECOG performance status of 0 - 2 (attachment 2)
* Life expectancy of at least 12 weeks
* At least 4 weeks since any prior surgery or radiotherapy. Patients who, in the opinion of the investigator, have fully recovered from surgery in less than 4 weeks may also be considered for the study. Patients must have recovered (CTC < 1) from acute toxicities of any previous therapy
* Granulocyte count > 1.5 x 109/L, platelet count > 100 x 109/L and hemoglobin >8.0 g/dL
* Serum bilirubin must be < 1.5 upper limit of normal (ULN) or ≤ 5 times ULN in patients with liver metastases. SGOT (AST) and SGPT (ALT) must be < 3 x ULN.
* Serum creatinine < 1.5 ULN or creatinine clearance > 60 ml/min
* Normal serum calcium
* Able to comply with study and follow-up procedures
* For all females of childbearing potential a negative pregnancy test must be obtained within 48 hours before registration starting therapy
* Patients with reproductive potential must use effective contraception
* Written (signed) Informed Consent to participate in the study.

Exclusion Criteria:

* Any unstable systemic disease [including active infection, uncontrolled hypertension, unstable angina, New York Heart Association (NYHA) Class III or IV heart failure (Attachment 3, NYHA Classification of Cardiac Disease), myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease] or Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
* Patients are excluded if they have brain metastasis or spinal cord compression that is newly diagnosed and/or has not yet been definitively treated with surgery and/or radiation; previously diagnosed and treated CNS metastases or spinal cord compression with evidence of stable disease (clinically stable imaging) for at least 2 months is permitted
* Any diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the study drug or that might affect the interpretation of the results or render the subject at high risk from treatment complications
* Nursing mothers
* Has known or suspected hypersensitivity or intolerance to boron, mannitol, or heparin, if an indwelling catheter is used
* Neuropathy ³ Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of VELCADE as determined by the rate of no progression at 6 weeks

SECONDARY OUTCOMES:
Efficacy of VELCADE as determined by
Objective response rate (incidence of CR and PR)
Disease control rate (CR, PR and stabilization)
Duration of disease control
Duration of objective response
Progression-free survival (PFS)
Overall survival (OS)
Safety of VELCADE
Rate of doublet therapy in second line

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles SORIA, MD, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France